CLINICAL TRIAL: NCT02234453
Title: A Phase 1 Trial Assessing the Safety and Performance of the Minicare H-2000 in Home Testing of Blood Counts in Chemotherapy Patients.
Brief Title: Home Testing of Blood Counts in Chemotherapy Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Leeds (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Principal Investigator, Dr Geoff Hall, Senior Lecturer & Honorary Consultant in Medical Oncology, University of Leeds
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MO14/11295
Record Dates: First submitted 2014-08-26; First posted 2014-09-09 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2016-06

CONDITIONS: Cancer
Keywords: cancer; chemotherapy; home; blood count; remote
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cancer patients (Experimental): Adult patients with solid tumours receiving systemic anti-cancer therapy who are able to use the Minicare H-2000.
  Interventions: Device: Minicare H-2000

INTERVENTIONS:
Device: Minicare H-2000 — Patients will use the Minicare H-2000 at home to measure their capillary blood count, temperature, record questionnaire results and transfer the results via the 3G network to the hospital team.

SUMMARY:
The investigators hypothesise that cancer patients on systemic anticancer therapy can measure a home blood count, temperature, record qualitative data and transfer the results electronically to the hospital clinical team.

A low neutrophil blood cell count (neutropenia) can be a dose-limiting toxicity of systemic anti-cancer therapy (SACT) and can be life-threatening when complicated by sepsis. Neutrophil count is usually obtained by venepuncture by a health-care professional. The Minicare H-2000 is a new device which facilitates home self-testing of blood count, temperature and symptoms. The four components are i) blood count recorder using a capillary sample obtained via finger-prick ii) Bluetooth linked thermometer iii) tele-hub collecting patient-reported outcomes and iv) secure communication through the 3G network.

The investigators propose a single-centre, non-randomised feasibility study to test the process of patients on chemotherapy using the Minicare H-2000 to deliver self-tested blood count readings, temperature and qualitative data electronically to the hospital clinical team. The aim is to test training of patients to use a finger-prick method of obtaining blood count, patient ability to perform the test, retention of training, the ability of the Minicare H-2000 to facilitate the data transfer and to test the secondary care interface. This study will provide preliminary data on the potential of Minicare H-2000 to prevent wasted hospital journeys when the blood count has not recovered sufficiently for subsequent SACT cycles. The investigators intend to obtain informed consent to recruit between 30 to 80 patients to this study which will be performed in addition to current local standard of care.

This study enables identification of suboptimal areas of the process prior to investigating the application of the minicare H-2000 within oncology to improve the clinical patient pathway. The investigators ongoing intentions are to trial the use of the Minicare H-2000 to reduce frequency and severity of neutropenic complications, prevent wasted hospital journeys and hospital resources, reduce non-elective hospital admissions and personalise delivery of SACT.

ELIGIBILITY:
Inclusion Criteria:

* Any solid tumour diagnosis being managed by either medical or clinical oncologists.
* Patients receiving one or more systemic chemotherapy drugs or targeted therapy at Leeds Cancer Centre.
* Adults ≥ 18 years.
* Live within boundaries of Local Care Direct service provision.
* Live in post-code with good 2G, 3G or GPRS connectivity according to coverage map.

Exclusion Criteria:

* On hormone treatment only for their cancer.
* Participating in the active phase of a therapeutic clinical trial.
* Inability to give informed consent due to mental capacity or language barrier.
* Patient or carer unable or unlikely to be able to perform fine manipulation required to use lancet or cartridge to obtain capillary blood sample and result.
* Known inherited or acquired bleeding disorder.
* History of haematological malignancy.
* Known poorly controlled anti-coagulation (INR>3.0 within 6 months)
* Prisoner in custody of HM Prison Service.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of home tested blood count results transferred to the hospital team on the day of the venous blood test performed prior to the subsequent SACT cycle | 15-42 days after training, dependent on length of chemotherapy cycle, most commonly 22 days.

SECONDARY OUTCOMES:
Proportion of home tested temperature and questionnaire responses transferred to the hospital after (i) initial home training (TP1), (ii) forty-eight hours (TP2) and (iii) on the day of venous blood test pre subsequent SACT cycle (TP3). | 15-42 days from training, dependent on length of chemotherapy cycle, most commonly 22 days.
Patient feedback on willingness to use and ease of use of Minicare H-2000. | 15 to 42 days
Assess proportion of successful tests performed with subsequent cycles. | up to 9 months. Most common maximum of 4.5 months.
Health-care professional feedback on server clinical interface. | 15-42 days, dependent on lenghtof chemotherapy cycle, most commonly 22 days.
Correlation of capillary granulocyte count with venous laboratory measured neutrophil count pre subsequent SACT cycle. | 15 to 42 days, dependent on chemotherapy cycle length, most commonly 22 days.
  Accuracy of the Minicare H-2000 granulocyte measuring technology will be confirmed using Pearson's correlation co-effcient and R squared.
Proportion of home tested blood count results transferred to the hospital team after (i) initial home training (TP1), (ii) forty-eight hours (TP2) | 24 to 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Geoff Hall, PhD, FRCP, Principal Investigator — University of Leeds
Locations (1):
- St James's Teaching Hospital, Leeds Teaching Hospitals NHS Trust, Leeds, West Yorkshire, United Kingdom